CLINICAL TRIAL: NCT05785780
Title: Optimizing Colorectal Cancer Screening Among Patients With Diabetes in Safety-Net Primary Care Settings: Targeting Implementation Approaches
Brief Title: Aim 3, Optimizing CRC Screening in Patients With Diabetes in Safety-net Primary Care Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Denalee O'Malley, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 002056; Pro2020002075 (Other: Rutgers, The State University of New Jersey); R00CA256043 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer Screening; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study uses a pilot, pre-post, hybrid effectiveness-implementation design to compare the adapted implementation strategy to usual care on: (1) effectiveness and (2) implementation outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted CRC Screening Toolkit (Experimental): Based on national survey data and a community engagement participatory implemention planning group, a tailored combination of widely accepted implementation strategies will be adapted for targeting CRC screening for patients with diabetes. These strategies include but are not limited to: identification of patient and practice-level barriers, patient education, provider reminders, and audit and feedback.
  Interventions: Behavioral: Targeted CRC Screening Toolkit

INTERVENTIONS:
Behavioral: Targeted CRC Screening Toolkit — Strategies in the toolkit include but are not limited to: identification of patient and practice-level barriers, routine tailored patient reminders, provider reminders, & clinic staff feedback.

SUMMARY:
This mixed methods study evaluates the effectiveness and feasibility of a multi-level (patient, team, organizations) intervention to optimize CRC screening for patients with diabetes in primary care safety-net settings.

DETAILED DESCRIPTION:
Aim 3 is a hybrid type 2 effectiveness-implementation pilot study in six primary care safety net clinics. This single-arm study uses a pre-post design to evaluate the targeted implementation strategies impact on: (1) preliminary effectiveness and (2) implementation (i.e., feasibility and acceptability) and a mixed-method comparative case study learning evaluation for safety-net primary care adoption and implementation. Implementation strategies that will be tested were developed through a stakeholder engaged, community-based participatory implementation planning approach. This study uses a tailored combination of implementation strategies that include but are not limited to: identification of patient and practice-level barriers, patient education matierals, patient reminders provider/clinical team education, clinical champions, and audit and feedback. The impact of this evaluation will be measure using mixed methods to assess Exploration, Preparation, Implementation factors related to how organizational and contextual variables affect adoption and implementation for targeting CRC screening among patients with diabetes in safety net clinics at 12 months post intervention. Aim 3 surveys 20 clinicians and staff from 6 clinics (n=120) and conducts key-informant interviews with 8 clinic and staff members at pre- and post-implementation (who have participated in the survey; n=96) and evaluates aggregate data for 30 patients across six clinics (n=180).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus;
* Participants not up-to-date with CRC screening based on electronic health record (e.g. FOBT/FIT in last year; flexible sigmoidoscopy within four years; or colonoscopy within nine years);
* Age-eligible for CRC screening (50-74 years of age);
* Participants in process of undergoing screening are eligible for participation if they have a FIT/FOBT incomplete test ordered for more than six months or a sigmoidoscopy or colonoscopy referral not completed for greater than one year.

Exclusion Criteria:

• Medical conditions not concordant with standard CRC screening intervals (e.g. prior CRC diagnosis, inflammatory bowel disease, renal failure, etc.).

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Colonoscopy uptake | 12 months
  Preliminary effectiveness: Clinic-level proportion of participants who complete a colonoscopy
Up-to-date CRC screening | 12 months
  Preliminary Effectiveness: Clinic-level proportion of participants who receive any CRC screening

SECONDARY OUTCOMES:
Rate of CRC Screening Uptake by Glucose Control (Controlled vs. Uncontrolled) Among Participants with Type 2 Diabetes | 12 months
  Preliminary Effectiveness: Clinic-level CRC screening by glucose control (controlled vs. uncontrolled)

OTHER OUTCOMES:
Participant Acceptability | 12 months
  Implementation: participants opt-out and non-adherence rates based on proportion of overall eligible participants
Implementation Fidelity | 12 months
  Clinic-level proportion of eligible participants who were contacted for screening based on implementation plan targets

CONTACTS AND LOCATIONS:
Overall Officials: Denalee O'Malley, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School; Rutgers Cancer Institute of New Jersey
Locations (1):
- RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Malley DM, Crabtree BF, Kaloth S, Ohman-Strickland P, Ferrante J, Hudson SV, Kinney AY. Strategic use of resources to enhance colorectal cancer screening for patients with diabetes (SURE: CRC4D) in federally qualified health centers: a protocol for hybrid type ii effectiveness-implementation trial. BMC Prim Care. 2024 Jul 5;25(1):242. doi: 10.1186/s12875-024-02496-0. PMID 38969987